CLINICAL TRIAL: NCT01644552
Title: Positive Angle Kappa: a Sign in Aniridia
Brief Title: Positive Angle Kappa
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1004M80112
Record Dates: First submitted 2012-02-20; First posted 2012-07-19 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Aniridia
Keywords: aniridia; positive angle kappa
MeSH Terms: conditions — Aniridia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- eye examinations

SUMMARY:
Patients with aniridia have positive angle kappas.

ELIGIBILITY:
Inclusion Criteria:

* patients with aniridia only

Exclusion Criteria:

* poor va
* PK,
* K-pro

Ages: 1 Month to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with aniridia
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Dept of ophthalmlogy, Minneapolis, Minnesota, United States